CLINICAL TRIAL: NCT02982083
Title: Clinical Trial on the Efficacy of Raloxifene on Disease Activity and Glucocorticoid-induced Osteoporosis in Postmenopausal Women With Rheumatoid Arthritis
Brief Title: Clinical Trial on the Efficacy of Raloxifene on Disease Activity in Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sara Saeidi Shahri (Other)
Responsible Party: Sponsor-Investigator, Sara Saeidi Shahri, Medical Student, Mashhad University of Medical Sciences
Organization: Mashhad University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 931755
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Raloxifene; Disease activity
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Raloxifene Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Evista (Active Comparator): 20 postmenopausal women suffering from rheumatoid arthritis that take raloxifene hydrochloride 60 mg oral tablets every day for one year.
  Interventions: Drug: Raloxifene hydrochloride
- Placebo (Placebo Comparator): 20 postmenopausal women suffering from rheumatoid arthritis that take placebo pills every day for one year.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Raloxifene hydrochloride — 20 patients consume raloxifene hydrochloride oral tablet daily for one year.
  Other Names: Evista
  Arms: Evista
Drug: Placebo Oral Tablet — 20 patients consume placebo oral tablets daily for one year.
  Arms: Placebo

SUMMARY:
The investigators select 40 postmenopausal women suffering from RA with 2.5<DAS28<5.5 referring to rheumatology clinics of Mashhad university of medical sciences and randomly divide them into intervention group and placebo group. Evista tab 60mg/day and placebo are administered double blind. In the beginning, total bone mineral density (BMD) assessment is carried out from all patients and then Alendronate is discontinued in 2 groups. In first 3 months, in addition to Evista and placebo, MTX tab 2.5mg is given to patients and they are allowed to consume NSAID with accurate record of its dosage. Patients visit rheumatologist monthly in these 3 months and NSAID should be discontinued 48 hours before every visit. At the end of month 3, disease activity and probable complications are evaluated and compared in 2 groups. Classic regimen should be started for every patient who doesn't enter remission phase in first 3 months.

In 4th month, DMARD regimen is administered and then patients are visited every 2 months. Clinical findings are collected in month 0, 1, 2, 3, 6, 8, 10, 12. After 12 months, another total BMD test is carried out and then data are analyzed including changes in BMD, DAS28, EULAR response criteria and HAQ-DI score.

ELIGIBILITY:
Inclusion Criteria:

* Patients are postmenopausal women.
* Patients should fit at least 4 criteria of ACR-1987 criteria for rheumatoid arthritis.
* Patients should be in range of 2.5 <DAS28-ESR <5.5

Exclusion Criteria:

* Patients with history of thrombotic events
* Patients suffering from another rheumatic diseases simultaneously
* Patients with sever symptoms of menopause
* Patients with known psychological diseases

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of DAS-28 criteria | 3 months
Assessing of complications | 3 months

SECONDARY OUTCOMES:
DAS-28 criteria | 12 months
Complications | 12 months
EULAR criteria | 12 months
HAQ-DI criteria | 12 months
Assessing of Bone Marrow Density score | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Sahebari, Professor, Study Director — Mashhad University of Medical Sciences

REFERENCES:
- [Derived] Sahebari M, Sarafraz Yazdi M, Mehrnaz Aghili S, Esmaily H, Saeidi S, Salari M. Efficacy of Raloxifene as Add-on Therapy on Disease Activity of Postmenopausal Women with Rheumatoid Arthritis: A Double-blind, Randomized, Placebo-controlled Clinical Trial. Curr Rheumatol Rev. 2023;19(1):93-101. doi: 10.2174/1573397118666220518114415. PMID 35585813